CLINICAL TRIAL: NCT06090019
Title: Effect of Self-Instructional Module Regarding Ventilator Associated Pneumonia Care Bundle Prevention on Internship Students' Knowledge and Clinical Performance in Pediatric Intensive Care Unit
Brief Title: Ventilator Associated Pneumonia Care Bundle Prevention on Internship Students' Knowledge and Clinical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAP
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Self-Instructional Module; Ventilator Associated Pneumonia; Care Bundle Prevention; Internship Students; Knowledge; Clinical Performance; Pediatric Intensive Care Unit
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Nursing interns students learned the routine nursing care of children on mechanically ventilation to prevent VAP by PICU nurses staff.
  Interventions: Behavioral: Routine PICU nursing care for children on mechanical ventilator.
- Study group (Experimental): Nursing interns students received comprehensive education about VAP care bundle prevention by self-instructional module through the researchers.
  Interventions: Behavioral: Self-instructional module for VAP care bundle prevention

INTERVENTIONS:
Behavioral: Routine PICU nursing care for children on mechanical ventilator. — Nursing interns students learned the routine PICU nursing care for the children on mechanical ventilator.
  Arms: Control group
Behavioral: Self-instructional module for VAP care bundle prevention — Nursing interns students learned about VAP care bundle prevention self-instructional module through assessment, preparation, implementation and evaluation phases.
  Arms: Study group

SUMMARY:
The goal of this clinical trial is to determine the effect of a self-instructional module regarding ventilator-associated pneumonia care bundle prevention on internship students' knowledge and clinical performance in pediatric intensive care unit.The hypotheses of this study were as follows:

1. Internship students who are taught by VAP care bundle prevention self-instructional module exhibit higher scores in knowledge test about VAP care bundle prevention than those who are not.
2. Internship students who are taught by VAP care bundle prevention self-instructional module exhibit higher scores in performing the VAP care bundle prevention procedure than those who are not.
3. Internship students who are taught by VAP care bundle prevention self-instructional module exhibit more positive feedback about it than those who are not.

ELIGIBILITY:
Inclusion Criteria:

* Nursing intern students at Faculty of Nursing, Alexandria university, Egypt.

Exclusion Criteria:

* No

Max Age: 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Nursing Interns' Knowledge | Before data collection, immediately after and after three months of the clinical experience
  total score ranged from 0 to 30 distributed as follows: Low knowledge level <60% of the total score, Moderate knowledge level from 60% to <75% of the total score, High knowledge level ≥75% of the total score.
Nursing Interns' performance | Before data collection, immediately after and after three months of the clinical experience
  Total score ranged from 16 to 32 and distributed as follows:
  Iow performance <60% of the total score, Moderate performance ranging from 60% to <75% of the total score, High performance for the score ≥75% of the total score.
Self-Instructional Module Feedback | immediately after VAP care bundle prevention self-instructional module
  It consists of 10 statements with 4 points Likert scale ranging from strongly disagree (1) to strongly agree (4). The higher score, the more positive feedback.

CONTACTS AND LOCATIONS:
Locations (1):
- Eman Arafa Badr, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abou Zed, S., & Mohammed, A. (2019). Impact of nursing guidelines on nurses' knowledge and performance regarding to prevention of ventilator-associated pneumonia in neonates. Journal of Nursing Education and Practice, 9(10), 1-14.
- [Background] Ali, S., & Elsayed, E. (2021). Effectiveness of self-instructional module on nurses' performance regarding caring of patient with acute respiratory distress during Covid-19 outbreaks. International Egyptian Journal of Nursing Sciences and Research, 2(2), 378-396. DOI: 10.21608/ejnsr.106256.1123.
- [Background] Antalova N, Klucka J, Rihova M, Polackova S, Pokorna A, Stourac P. Ventilator-Associated Pneumonia Prevention in Pediatric Patients: Narrative Review. Children (Basel). 2022 Oct 9;9(10):1540. doi: 10.3390/children9101540. PMID 36291475
- [Background] Benito, S., Bantulo, S., Haudar, F. (2022). Effectiveness of Self Learning Modules in Teaching Mathematcs. Journal of Recent Research in Thesis and Dissertation (IJRRTD) Vol. 3(1), pp: (33-45)DOI: https://doi.org/10.5281/zenodo.6497186 Available at: www.paperpublications.org
- [Background] Dsilva, F., Mathew, S., & Gincy, J. (2022). Effectiveness of a self-instructional module on knowledge and observed practices of nurses with regard to prevention of central line-associated blood stream infection. A Before-After Intervention Study Journal of Health Management, 24(2), 233-239,